CLINICAL TRIAL: NCT00000475
Title: Prevention of Early Readmission in Elderly Congestive Heart Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 64; R29HL044739 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure

INTERVENTIONS:
Behavioral: health education

SUMMARY:
To assess the impact of a multidisciplinary treatment program on three-month readmission-free survival in elderly congestive heart failure patients.

DETAILED DESCRIPTION:
BACKGROUND:

The prevalence of congestive heart failure increases progressively with advancing age, and congestive heart failure is a major cause of mortality, morbidity, and diminished quality of life in the elderly. Not only is congestive heart failure the most common cardiovascular indication for hospitalization in patients 65 years or older, but frequent repetitive hospitalizations, occurring in 30-50 percent of patients within three to six months of initial discharge, create an imposing cost burden in caring for these patients. A pilot study conducted at the grantee institution has shown that elderly congestive heart failure patients at risk for early readmission can be identified at the time of initial hospitalization, that up to 50 percent of readmissions are potentially preventable, and that a non-pharmacologic treatment strategy consisting of patient education, medication analysis, discharge planning, and enhanced follow-up is feasible and may reduce readmissions by 30 to 50 percent.

DESIGN NARRATIVE:

In the feasibility study, patients were randomly assigned to receive intervention or standard care over a four year period. Patients were stratified into readmission risk categories of high or moderate based on the presence of four independent risk factors for readmission defined in a prior study at Jewish Hospital in St. Louis. The risk factors included: four or more prior hospitalizations within the preceding five-year interval, previous history of congestive heart failure, hypocholesterolemia, and right bundle-branch block on the admitting electrocardiogram. The study intervention consisted of individualized patient education using teaching materials specifically designed for the study; a careful review of medications with specific recommendations designed to eliminate unnecessary drugs, decrease the number of dosing intervals, improve compliance, and minimize side effects; early discharge planning; and enhanced post-discharge follow-up. The primary endpoints were rehospitalization within 90 days after initial hospital discharge and the cumulative number of days hospitalized during follow-up. Principal secondary endpoints included analyses of the effect of the study intervention on compliance with prescribed medications, dietary sodium intake, incidence of adverse drug reactions, patient knowledge and understanding of congestive heart failure, patient-assessed quality of life, and the overall cost of medical care.

In the full-scale trial, 140 patients were assigned to the control group which received all standard treatments and services ordered by their physicians. A total of 142 patients were assigned to the treatment group which received intensive education about congestive heart failure and its treatment by an experienced cardiovascular research nurse, using a teaching booklet developed by study investigators for geriatric patients with heart failure. Treatment group patients also received individualized dietary assessment and instruction given by a registered dietitian; consultation with social-service personnel to facilitate discharge planning and care after discharge; an analysis of medications by a geriatric cardiologist who made specific recommendations to eliminate unnecessary medications and simplify the overall regimen; and intensive follow-up after discharge. The goals of follow-up were to reinforce the patient's education, ensure compliance with medications and diet, and identify recurrent symptoms amenable to treatment on an outpatient basis. The primary outcome measure was survival for 90 days without hospital readmission. Secondary endpoints included the number of readmissions for any cause, the number of readmissions for congestive heart failure, the cumulative number of days of hospitalization during follow-up, quality-of-life scores, and the overall cost of medical care.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Men and women, ages 70 or older, with documented congestive heart failure.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1990-04; Study Completion 1995-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rich — Jewish Hospital and St. Mary's Healthcare

REFERENCES:
- [Background] Rich MW, Beckham V, Wittenberg C, Leven CL, Freedland KE, Carney RM. A multidisciplinary intervention to prevent the readmission of elderly patients with congestive heart failure. N Engl J Med. 1995 Nov 2;333(18):1190-5. doi: 10.1056/NEJM199511023331806. PMID 7565975
- [Background] Rich MW, Vinson JM, Sperry JC, Shah AS, Spinner LR, Chung MK, Davila-Roman V. Prevention of readmission in elderly patients with congestive heart failure: results of a prospective, randomized pilot study. J Gen Intern Med. 1993 Nov;8(11):585-90. doi: 10.1007/BF02599709. PMID 8289096